CLINICAL TRIAL: NCT01645202
Title: A Randomized Comparison of Transcatheter Heart Valves in High Risk Patients With Severe Aortic Stenosis: Medtronic CoreValve Versus Edwards SAPIEN XT (The CHOICE Trial)
Brief Title: A Comparison of Transcatheter Heart Valves in High Risk Patients With Severe Aortic Stenosis: The CHOICE Trial
Acronym: CHOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Segeberger Kliniken GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SK 107 -- 012/12 (II)
Record Dates: First submitted 2012-06-06; First posted 2012-07-20 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-02

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; TAVI; Device success; Aortic regurgitation
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAVI with Edwards Sapien XT valve (Active Comparator)
  Interventions: Procedure: Transcatheter Aortic Valve Implantation (TAVI)
- TAVI with Medtronic CoreValve (Active Comparator)
  Interventions: Procedure: Transcatheter Aortic Valve Implantation (TAVI)

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Implantation (TAVI) — Comparison of different types of valves
  Other Names: Transcatheter Aortic Valve Replacement (TAVR)

SUMMARY:
A randomized controlled multicenter study comparing the acute hemodynamic performance of the Edwards Sapien XT and the Medtronic CoreValve transcatheter heart valves in high risk patients with severe symptomatic aortic stenosis.

DETAILED DESCRIPTION:
Study design: randomized open-label multicenter

Primary endpoint:

'Device success' as recently defined by VARC which is a 'technical' composite endpoint including:

1. Successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system,
2. Correct position of the device in the proper anatomical location,
3. Intended performance of the prosthetic heart valve (aortic valve area > 1.2 cm2 and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, without moderate or severe prosthetic valve AR) and
4. Only one valve implanted in the proper anatomical location.

Secondary endpoints:

* 30-day-combined safety endpoint which is a combined endpoint defined by VARC as:

  1. All cause mortality,
  2. Major stroke,
  3. Life threatening (or disabling) bleeding,
  4. Acute kidney injury-Stage 3 (including renal replacement therapy),
  5. Periprocedural myocardial infarction,
  6. Major vascular complications and
  7. Repeat procedure for valve-related dysfunction (surgical or interventional therapy). *
* Combined efficacy endpoint at 1 year which is a composite endpoint defined by VARC as:

  1. All cause mortality between 30 days and one year,
  2. Failure of current therapy for aortic stenosis, requiring hospitalization for symptoms of valve-related or cardiac decompensation and
  3. Prosthetic heart valve dysfunction (aortic valve area < 1.2 cm2 and mean aortic valve gradient > 20 mmHg or peak velocity > 3 m/s or moderate or severe prosthetic valve AR). *
* Cardiovascular mortality as defined by VARC at 1 month, 6 and 12 months. *
* Major adverse cardiovascular and cerebrovascular events (MACCE): myocardial infarction, cardiac or vascular surgery and stroke at 30 days, 6 & 12 months.
* Rehospitalization for heart failure at 12 months
* Quality of life (assessed with the Euro5Qual-questionnaire) at 12 months
* NYHA-class improvement at 30 days, 6 and 12 months
* Vascular complication as defined by VARC at 30 days.
* Post-procedural pacemaker implantation at 1 month
* Major or minor Bleeding at 30 days as defined be VARC.

ELIGIBILITY:
Inclusion Criteria:

1. Severe aortic valve stenosis defined as aortic valve area (AVA) ≤ 1cm2 or 0.6 cm2/m2
2. Presence of clinical symptoms defined as New York Heart Association (NYHA) functional class ≥ 2
3. Age > 75 years and/or Logistic EuroSCORE ≥ 20% and/or STS risk score ≥ 10% and/or contraindication to conventional surgical aortic valve replacement (porcelain aorta, previous chest radiation, chest deformation)
4. Native aortic valve annulus measuring 20-25 mm
5. Patients must be suitable for a transfemoral vascular access
6. The patient signing a written informed consent prior to intervention

Exclusion Criteria:

1. Life expectancy < 12 months due to co-morbid conditions
2. Native aortic valve annulus < 20 mm and > 25 mm (this could be amended if further valve sizes for the transfemoral approach become available for both prostheses during the study period)
3. Pre-existing aortic bioprosthesis
4. Cardiogenic shock or hemodynamic instability
5. History of, or active endocarditis
6. Contraindications for a transfemoral access
7. Active peptic ulcer or upper gastro-intestinal bleeding within the prior 3 months.
8. Hypersensitivity or contraindication to aspirin, heparin or clopidogrel
9. Active infection requiring antibiotic treatment
10. An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 3 months post-enrolment
11. Patients actively participating in another drug or device investigational study and have not yet completed the primary endpoint follow-up period

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 241 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
'Device success' as recently defined by the Valve Academic Research Consortium | Immediately after the procedure
  Device success is a 'technical' composite endpoint including successful vascular access, delivery and deployment of the device and successful retrieval of the delivery system, correct position of the device in the proper anatomical location, intended performance of the prosthetic heart valve (aortic valve area > 1.2 cm2 and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, without moderate or severe prosthetic valve AR) and only one valve implanted in the proper anatomical location.

SECONDARY OUTCOMES:
VARC-defined combined safety endpoint | 30 days
  Combined endpoint defined by VARC as: 1) All cause mortality, 2) Major stroke, 3) Life threatening (or disabling) bleeding, 4) Acute kidney injury-Stage 3 (including renal replacement therapy), 5) Periprocedural myocardial infarction, 6) Major vascular complications and 7) Repeat procedure for valve-related dysfunction (surgical or interventional therapy).
VARC-defined combined efficacy endpoint | 1 year
  A composite endpoint defined by VARC as: 1) All cause mortality between 30 days and one year, 2) Failure of current therapy for aortic stenosis, requiring hospitalization for symptoms of valve-related or cardiac decompensation and 3) Prosthetic heart valve dysfunction (aortic valve area < 1.2 cm2 and mean aortic valve gradient > 20 mmHg or peak velocity > 3 m/s or moderate or severe prosthetic valve AR)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdel-Wahab, MD, Principal Investigator — Herzzentrum, Segeberger Kliniken, Bad Segeberg, Germany; Gert Richardt, MD, Study Chair — Herzzentrum, Segeberger Kliniken, Bad Segeberg, Germany
Locations (1):
- Segeberger Kliniken GmbH / Herzzentrum, Bad Segeberg, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Brown DL, Block PC, Guyton RA, Pichard AD, Bavaria JE, Herrmann HC, Douglas PS, Petersen JL, Akin JJ, Anderson WN, Wang D, Pocock S; PARTNER Trial Investigators. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Engl J Med. 2010 Oct 21;363(17):1597-607. doi: 10.1056/NEJMoa1008232. Epub 2010 Sep 22. PMID 20961243
- [Background] Grube E, Schuler G, Buellesfeld L, Gerckens U, Linke A, Wenaweser P, Sauren B, Mohr FW, Walther T, Zickmann B, Iversen S, Felderhoff T, Cartier R, Bonan R. Percutaneous aortic valve replacement for severe aortic stenosis in high-risk patients using the second- and current third-generation self-expanding CoreValve prosthesis: device success and 30-day clinical outcome. J Am Coll Cardiol. 2007 Jul 3;50(1):69-76. doi: 10.1016/j.jacc.2007.04.047. Epub 2007 Jun 6. PMID 17601548
- [Background] Moat NE, Ludman P, de Belder MA, Bridgewater B, Cunningham AD, Young CP, Thomas M, Kovac J, Spyt T, MacCarthy PA, Wendler O, Hildick-Smith D, Davies SW, Trivedi U, Blackman DJ, Levy RD, Brecker SJ, Baumbach A, Daniel T, Gray H, Mullen MJ. Long-term outcomes after transcatheter aortic valve implantation in high-risk patients with severe aortic stenosis: the U.K. TAVI (United Kingdom Transcatheter Aortic Valve Implantation) Registry. J Am Coll Cardiol. 2011 Nov 8;58(20):2130-8. doi: 10.1016/j.jacc.2011.08.050. Epub 2011 Oct 20. PMID 22019110
- [Background] Abdel-Wahab M, Zahn R, Horack M, Gerckens U, Schuler G, Sievert H, Eggebrecht H, Senges J, Richardt G; German transcatheter aortic valve interventions registry investigators. Aortic regurgitation after transcatheter aortic valve implantation: incidence and early outcome. Results from the German transcatheter aortic valve interventions registry. Heart. 2011 Jun;97(11):899-906. doi: 10.1136/hrt.2010.217158. Epub 2011 Mar 12. PMID 21398694
- [Background] Sherif MA, Abdel-Wahab M, Stocker B, Geist V, Richardt D, Tolg R, Richardt G. Anatomic and procedural predictors of paravalvular aortic regurgitation after implantation of the Medtronic CoreValve bioprosthesis. J Am Coll Cardiol. 2010 Nov 9;56(20):1623-9. doi: 10.1016/j.jacc.2010.06.035. PMID 21050971
- [Derived] Abdel-Wahab M, Landt M, Neumann FJ, Massberg S, Frerker C, Kurz T, Kaur J, Toelg R, Sachse S, Jochheim D, Schafer U, El-Mawardy M, Robinson DR, Richardt G; CHOICE Investigators. 5-Year Outcomes After TAVR With Balloon-Expandable Versus Self-Expanding Valves: Results From the CHOICE Randomized Clinical Trial. JACC Cardiovasc Interv. 2020 May 11;13(9):1071-1082. doi: 10.1016/j.jcin.2019.12.026. Epub 2020 Apr 15. PMID 32305398
- [Derived] Abdel-Wahab M, Neumann FJ, Mehilli J, Frerker C, Richardt D, Landt M, Jose J, Toelg R, Kuck KH, Massberg S, Robinson DR, El-Mawardy M, Richardt G; CHOICE Investigators. 1-Year Outcomes After Transcatheter Aortic Valve Replacement With Balloon-Expandable Versus Self-Expandable Valves: Results From the CHOICE Randomized Clinical Trial. J Am Coll Cardiol. 2015 Aug 18;66(7):791-800. doi: 10.1016/j.jacc.2015.06.026. PMID 26271061
- [Derived] Abdel-Wahab M, Mehilli J, Frerker C, Neumann FJ, Kurz T, Tolg R, Zachow D, Guerra E, Massberg S, Schafer U, El-Mawardy M, Richardt G; CHOICE investigators. Comparison of balloon-expandable vs self-expandable valves in patients undergoing transcatheter aortic valve replacement: the CHOICE randomized clinical trial. JAMA. 2014 Apr 16;311(15):1503-14. doi: 10.1001/jama.2014.3316. PMID 24682026